CLINICAL TRIAL: NCT02150967
Title: A Phase II Multicenter, Single Arm Study of Oral BGJ398 in Adult Patients With Advanced or Metastatic Cholangiocarcinoma With FGFR2 Gene Fusions or Other FGFR Genetic Alterations Who Failed or Are Intolerant to Platinum-based Chemotherapy
Brief Title: A Phase II, Single Arm Study of BGJ398 in Patients With Advanced Cholangiocarcinoma
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was terminated early due to limited efficacy in Cohorts 2 and 3 (exploratory endpoints). Termination was not due to concerns about safety and had no impact on the primary efficacy analysis (ie, results reported for Cohort 1).
Sponsor: QED Therapeutics, a BridgeBio company (Industry)
Collaborators: Helsinn Healthcare SA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CBGJ398X2204; 2013-005085-19 (EudraCT Number)
Record Dates: First submitted 2014-05-12; First posted 2014-05-30 (Estimated); Results first posted 2022-07-15 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Advanced Cholangiocarcinoma; FGFR2 Gene Mutation
Keywords: cholangiocarcinoma,; FGFR2 gene fusion,; FGFR genetic alteration
MeSH Terms: conditions — Cholangiocarcinoma | interventions — infigratinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- BGJ398 (infigratinib) (Experimental): To estimate the anti-tumor activity of BGJ398 (infigratinib)
  Interventions: Drug: BGJ398 (infigratinib)

INTERVENTIONS:
Drug: BGJ398 (infigratinib) — Capsule for oral use

SUMMARY:
This is a multi-center, open label, single arm phase II study evaluating BGJ398 (infigratinib) anti-tumor activity in advanced or metastatic cholangiocarcinoma patients with fibroblast growth factor receptor (FGFR) genetic alterations.

DETAILED DESCRIPTION:
Adult patients with histologically or cytologically confirmed advanced or metastatic cholangiocarcinoma with FGFR2 gene fusions or translocations or other FGFR genetic alterations have been enrolled. Subjects must have received at least one prior regimen containing gemcitabine with or without cisplatin for advanced/metastatic disease. Subjects should have had evidence of progressive disease following their prior regimen or if prior treatment was discontinued due to toxicity must have continued evidence of measurable disease. Up to approximately 160 adult patients over age 18, both male and female were planned for enrollment.

Three cohorts of subjects comprise the study population:

Cohort 1: subjects with FGFR2 gene fusions (ie, fusions or rearrangements [formerly translocations]).

Cohort 2: subjects with FGFR genetic alterations other than FGFR2 gene fusions or rearrangements.

Cohort 3: subjects with FGFR2 gene fusions or rearrangements who have received a prior FGFR inhibitor.

All subjects received oral BGJ398 (infigratinib), once-daily, on a three weeks on (21 days), one week off (7 days) schedule. One treatment cycle consists of 28 days.

Notes:

Cohort 1 was pre-specified as the primary analysis population. Results of these analyses were previously disclosed (posted 22 June 2022). There were no additional efficacy or safety endpoints to assess in Cohort 1 after primary completion (01 March 2021).

Cohorts 2 and 3 were added at protocol amendment (PA) 4 to support only exploratory efficacy objectives of the study. These cohorts were ongoing the time of primary completion (01 March 2021). After interim review of the data from these cohorts (as permitted by the protocol) only limited efficacy was observed and the sponsor terminated the study early. Therefore, a formal efficacy analysis was not performed for Cohorts 2 and 3. However, baseline characteristics and safety data were analyzed.

ELIGIBILITY:
Inclusion criteria:

- Adult patients with histologically or cytologically confirmed cholangiocarcinoma at the time of diagnosis.

Patients with cancers of the gallbladder or ampulla of Vater are not eligible.

- Patients must have received at least one prior regimen containing gemcitabine with or without cisplatin for advanced/ metastatic disease. Patient should have evidence of progressive disease following prior regimen, or if prior treatment discontinued due to toxicity must have continued evidence of measurable or evaluable disease.

Exclusion criteria:

* Prior or current treatment with a MEK inhibitor (all Cohorts), BGJ398 (infigratinib) (all Cohorts), or selective FGFR inhibitor (Cohorts 1 and 2 only).
* insufficient organ function

  * Absolute Neutrophil Count (ANC) < 1,000/mm3 [1.0 x 10^9/L]
  * Platelets < 75,000/mm3 [75 x 10^9/L]
  * Hemoglobin < 109.0 g/dL
  * Total bilirubin > 1.5x upper limit of normal (ULN)
  * Aspartate aminotransferase/glutamic oxaloacetic transaminase (AST/SGOT) and alanine aminotransferase/glutamic pyruvic transaminase (ALT/SGPT) > 2.5x ULN (AST and ALT > 5x ULN in the presence of liver metastases)
  * Serum creatinine > 1.5x ULN and a calculated or measured creatinine clearance < 45 mL/min
  * Inorganic phosphorus outside of normal limits
  * Total and ionized serum calcium outside of normal limits

Other protocol-defined inclusion/exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 143 (Actual)
Dates: Start 2014-07-23 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2022-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: QED Therapeutics, Study Director — QED Therapeutics
Locations (30):
- United States (8):
  - QED Investigative Site, Phoenix, Arizona
  - QED Investigative Site, Los Angeles, California
  - QED Investigative Site, San Francisco, California
  - QED Investigative Site, Boston, Massachusetts
  - QED Investigative Site, Detroit, Michigan
  - QED Investigative Site, New York, New York
  - QED Investigative Site, Columbus, Ohio
  - QED Investigative Site, Houston, Texas
- Belgium (2):
  - QED Investigative Site, Brussels
  - QED Investigative Site, Leuven
- Germany (3):
  - QED Investigative Site, Cologne, North Rhine-Westphalia
  - QED Investigative Site, Heidelberg
  - QED Investigative Site, Tübingen
- Italy (3):
  - QED Investigative Site, Ancona, AN
  - QED Investigative Site, Milan, MI
  - QED Investigative Site, Roma, RM
- Russia (2):
  - QED Investigative Site, Moscow
  - QED Investigative Site, Volzhskiy
- QED Investigative Site, Singapore, Singapore
- QED Investigative Site, Seoul, Korea, South Korea
- Spain (2):
  - QED Investigative Site, Barcelona
  - QED Investigative Site, Madrid
- Taiwan (2):
  - QED Investigative Site, Taipei, Taiwan ROC
  - QED Investigative Site, Zhunan
- Thailand (2):
  - QED Investigative Site, Khon Kaen, THA
  - QED Investigative Site, Bangkok
- United Kingdom (4):
  - QED Investigative Site, Bebington
  - QED Investigative Site, Birmingham
  - QED Investigative Site, Manchester
  - QED Investigative Site, Nottingham

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Javle M, Roychowdhury S, Kelley RK, Sadeghi S, Macarulla T, Weiss KH, Waldschmidt DT, Goyal L, Borbath I, El-Khoueiry A, Borad MJ, Yong WP, Philip PA, Bitzer M, Tanasanvimon S, Li A, Pande A, Soifer HS, Shepherd SP, Moran S, Zhu AX, Bekaii-Saab TS, Abou-Alfa GK. Infigratinib (BGJ398) in previously treated patients with advanced or metastatic cholangiocarcinoma with FGFR2 fusions or rearrangements: mature results from a multicentre, open-label, single-arm, phase 2 study. Lancet Gastroenterol Hepatol. 2021 Oct;6(10):803-815. doi: 10.1016/S2468-1253(21)00196-5. Epub 2021 Aug 3. PMID 34358484
- [Derived] Javle M, Lowery M, Shroff RT, Weiss KH, Springfeld C, Borad MJ, Ramanathan RK, Goyal L, Sadeghi S, Macarulla T, El-Khoueiry A, Kelley RK, Borbath I, Choo SP, Oh DY, Philip PA, Chen LT, Reungwetwattana T, Van Cutsem E, Yeh KH, Ciombor K, Finn RS, Patel A, Sen S, Porter D, Isaacs R, Zhu AX, Abou-Alfa GK, Bekaii-Saab T. Phase II Study of BGJ398 in Patients With FGFR-Altered Advanced Cholangiocarcinoma. J Clin Oncol. 2018 Jan 20;36(3):276-282. doi: 10.1200/JCO.2017.75.5009. Epub 2017 Nov 28. PMID 29182496
- [Derived] Borad MJ, Gores GJ, Roberts LR. Fibroblast growth factor receptor 2 fusions as a target for treating cholangiocarcinoma. Curr Opin Gastroenterol. 2015 May;31(3):264-8. doi: 10.1097/MOG.0000000000000171. PMID 25763789

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with a diagnosis of advanced or metastatic cholangiocarcinoma were recruited to this open-label, single-arm global study across 20 centers (9 in the US, 5 in W. Europe, 6 in Asia) based on documented evidence of FGFR gene alteration. The first participant was treated on 23 July 2014. The data cutoff for the primary analysis (Cohort 1 only) was 01 March 2021.The data cutoff for the final analysis (Cohort 2 and 3 only) was 07 February 2022.
Pre-assignment Details: Subjects meeting inclusion/exclusion criteria were enrolled into the following cohorts:
  Cohort 1 (FGFR2 fusions): Primary analysis population (N=108). Cohort 2 (Other FGFR alterations): N=25. Cohort 3 (FGFR2 fusions and prior FGFR inhibitor): N=10.
  Note:
  Primary efficacy outcome measures were prespecified only for Cohort 1. Cohorts 2 and 3 were added following PA 4 to support exploratory objectives only.
  Cohorts 2 and 3 are not the primary analysis population.
Groups:
- Cohort 1: FGFR2 Fusions; Cohort 2: Other FGFR Alterations; Cohort 3: FGFR2 Fusions and Prior FGFR Inhibitor: Infigratinib 125 mg once daily (3 wk on/1 wk off treatment)
Period: Overall Study
Arm/Group | Cohort 1: FGFR2 Fusions | Cohort 2: Other FGFR Alterations | Cohort 3: FGFR2 Fusions and Prior FGFR Inhibitor
Started | 108 | 25 | 10
Treatment Ongoing | 0 | 0 | 0
Treatment Ended (Per protocol, patients continue treatment until radiographical documentation of disease progression.) | 108 | 25 | 10
Completed (Cohort 1: completed is defined as patients who had the opportunity to be followed for at least 10 months after their initial exposure of infigratinib. This cohort supports the primary efficacy analysis of the study Cohort 2 and 3: completed is defined as patients who may have had the opportunity to be followed for at least 10 months after their initial exposure of infigratinib or up to the time of study termination. These cohorts support only the exploratory endpoints of the study) | 108 (Cohort 1 (FGFR2 fusions): Primary efficacy outcome measures were prespecified only for this cohort.) | 25 (Cohort 2 (Other FGFR Alterations): not the primary efficacy analysis population.) | 10 (Cohort 3 (FGFR2 fusions and prior FGFR inhibitor): not the primary efficacy analysis population.)
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS), defined as all subjects who had received at least 1 dose of infigratinib.
Groups:
- Cohort 2: Other FGFR Genetic Alterations; Cohort 3: FGFR2 Fusions and Prior FGFR Inhibitor: Infigratinib 125 mg once daily (3 wk on/1 wk off treatment)
- Total: Total of all reporting groups
Arm/Group | Cohort 1: FGFR2 Fusions | Cohort 2: Other FGFR Genetic Alterations | Cohort 3: FGFR2 Fusions and Prior FGFR Inhibitor | Total
Number analyzed (Participants) | 108 | 25 | 10 | 143
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 82 | 17 | 8 | 107
  >=65 years | 26 | 8 | 2 | 36
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.4 (13.08) | 59.9 (9.89) | 51.8 (12.07) | 54.0 (12.88)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 67 | 12 | 3 | 82
  Male | 41 | 13 | 7 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 11 | 2 | 0 | 13
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 4 | 1 | 2 | 7
  White | 78 | 22 | 8 | 108
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 15 | 0 | 0 | 15
Region of Enrollment [Count of Participants; unit: Participants]
  North America | 77 | 12 | 5 | 94
  Europe | 24 | 11 | 5 | 40
  South Korea | 0 | 1 | 0 | 1
  Singapore | 4 | 0 | 0 | 4
  Taiwan | 1 | 0 | 0 | 1
  Thailand | 2 | 1 | 0 | 3
ECOG PS [Count of Participants; unit: Participants] — Functional status was assessed at baseline using the Eastern Cooperative Oncology Group Performance Scale (ECOG PS), defined as follows:
  0. Fully active, able to carry out all pre-disease performance without restriction.
  1. Restricted in physically strenuous activity but ambulatory and able to carry out work of a light or sedentary nature.
  2. Ambulatory and capable of all selfcare but unable to carry out any work activities; up and about more than 50% of waking hours.
  3. Capable of only limited selfcare; confined to bed or chair more than 50% of waking hours.
  4. Completely disabled.
  Participants
    0 | 45 | 11 | 3 | 59
    1 | 62 | 13 | 7 | 82
    2 | 1 | 1 | 0 | 2
Primary site of cancer [Count of Participants; unit: Participants]
  Bile Duct | 105 | 24 | 10 | 139
  Cholangiocarcinoma | 1 | 1 | 0 | 2
  Liver | 2 | 0 | 0 | 2
Non-Liver Metastatic Site [Count of Participants; unit: Participants]
  No metastatic site | 5 | 4 | 0 | 9
  Had metastatic site | 102 | 21 | 10 | 133
  Missing | 1 | 0 | 0 | 1
Non-Liver Metastatic Site [Count of Participants; unit: Participants] — Data represent the number of patients in the FAS with at least one metastatic site. Note that for some patients, metastases may have been reported at more than one site.
  Participants
    Bone | 28 | 1 | 2 | 31
    Lung | 74 | 9 | 2 | 85
    Node | 62 | 5 | 1 | 68
    Other | 41 | 6 | 2 | 49
Time from initial diagnosis to first dose day [Median (Full Range); unit: months] | 12.75 [1.74 to 152.94] | 16.49 [5.62 to 176.59] | 22.11 [11.86 to 61.80] | 15 [1.74 to 176.59]
Time from the most recent recurrence/progression to the first dose day [Median (Full Range); unit: months] — Population: The date of most recent recurrence/progression is based on medical history which may not have been available for all patients.
  months
    number analyzed (Participants) | 98 | 23 | 10 | 131
    (all) | 1.40 [0.03 to 14.59] | 1.31 [0.30 to 8.28] | 1.36 [0.49 to 13.74] | 1.36 [0.03 to 14.59]
Histological Grade [Count of Participants; unit: Participants]
  Well differentiated | 9 | 2 | 0 | 11
  Moderately differentiated | 42 | 14 | 7 | 63
  Poorly differentiated | 33 | 2 | 2 | 37
  Undifferentiated | 1 | 0 | 0 | 1
  Unknown/missing | 22 | 7 | 1 | 30
  Not Applicable | 1 | 0 | 0 | 1
Stage at Time of Study Entry [Count of Participants; unit: Participants] — The AJCC staging manual (7th edition) for intrahepatic cholangiocarcinoma was used for cancer staging at baseline, defined as follows:
  Stage I: solitary tumor without vascular invasion. Stage II: solitary tumor with vascular invasion or multiple tumors with or without vascular invasion.
  Stage III: tumor perforating the visceral peritoneum or involving local hepatic structure by direct invasion.
  Stage IV: tumor with periductal invasion, or any tumor with regional lymph node metastasis present, or any tumor with or without lymph node metastasis but metastasized to a distant site.
  Participants
    Stage II | 1 | 3 | 0 | 4
    Stage III | 0 | 2 | 0 | 2
    Stage IV | 107 | 20 | 10 | 137

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR) as Assessed by Blinded Independent Central Imaging Review (BICR)
Description: ORR is defined as the percentage (%) of subjects with a best overall response of Complete Response (CR) or Partial Response (PR), as per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1, evaluated by computed tomography (CT) or magnetic resonance imaging (MRI) scans every 28 days.
  RECIST (v1.1) response criteria were as follows:
  CR: disappearance of all target lesions. Any pathological lymph node (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease from baseline in the sum of diameters of all target lesions.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (FGFR fusions). Results were previously disclosed (22 June 2022). There are no additional efficacy endpoints to assess for Cohort 1, thus efficacy data were not re-analyzed for the final analysis.
  Due to early termination of the study, no formal efficacy analyses were performed for Cohorts 2 and 3.
Time Frame: Analysis was conducted when all subjects in Cohort 1 had the opportunity to be followed for at least 10 months after their initial exposure to infigratinib. Data cutoff 01 March 2021.
Population: Full Analysis Set (FAS), defined as all subjects in Cohort 1 who had received at least one dose of infigratinib.
Measure: Number (95% Confidence Interval); unit: Percentage (%) of subjects with CR or PR
Arm/Group | Cohort 1: FGFR2 Fusions
Number analyzed (Participants) | 108
Percentage (%) of subjects with CR or PR | 23.1 [15.6 to 32.2]

2. Secondary Outcome: Overall Response Rate (ORR) as Assessed by the Investigator
Description: ORR is defined as the percentage (%) of subjects with a best overall response of CR or PR, evaluated by CT or MRI scans every 28 days.
  RECIST (v1.1) response criteria were as follows:
  CR: disappearance of all target lesions. Any pathological lymph node (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease from baseline in the sum of diameters of all target lesions.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (FGFR fusions) only. These results were previously disclosed (22 June 2022).
  There are no additional efficacy endpoints to assess for Cohort 1, thus efficacy data were not re-analyzed for the final analysis.
  Due to early termination of the study, no formal efficacy analyses were performed for Cohorts 2 and 3.
Time Frame: Analysis conducted when all subjects in Cohort 1 had the opportunity to be followed for at least 10 months after their initial exposure to infigratinib. Data cutoff for the primary analysis was 01 March 2021.
Population: Full Analysis Set (FAS), defined as all subjects in Cohort 1 who had received at least one dose of infigratinib.
Measure: Number (95% Confidence Interval); unit: Percentage (%) of subjects with CR or PR
Groups:
- Cohort 1: FGFR2 Fusion/Rearrangements: Infigratinib 125 mg once daily (3 wk on/1 wk off treatment)
Arm/Group | Cohort 1: FGFR2 Fusion/Rearrangements
Number analyzed (Participants) | 108
Percentage (%) of subjects with CR or PR | 32.4 [23.7 to 42.1]

3. Secondary Outcome: Best Overall Response (BOR)
Description: BOR is defined as the best overall response a subject achieved during the study before any subsequent antineoplastic therapy. The endpoint is summarized for the rate of BOR of CR, PR, progressive disease (PD), and stable disease (SD), evaluated by CT or MRI scans every 28 days.
  RECIST (v1.1) response criteria were as follows:
  CR: disappearance of all target lesions. Any pathological lymph node (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease from baseline in the sum of diameters of all target lesions.
  PD: at least a 20% increase in the sum of diameters of all target lesions from that of the smallest sum on study and an absolute increase in target lesion of at least 5mm.
  SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (FGFR fusion)
Time Frame: Analysis conducted when all subjects in Cohort 1 had the opportunity to be followed for at least 10 months after their initial exposure to infigratinib. Data cutoff 01 March 2021.
Population: Full Analysis Set (FAS), defined as all subjects in Cohort 1 who had received at least one dose of infigratinib.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: FGFR2 Fusion/Rearrangements
Number analyzed (Participants) | 108
Participants
  BOR by BICR: Confirmed CR | 1
  BOR by BICR: Confirmed PR | 24
  BOR by BICR: Stable Disease | 66
  BOR by BICR: Progressive Disease | 11
  BOR by BICR: Not Done | 6
  BOR by Investigator: Confirmed CR | 0
  BOR by Investigator: Confirmed PR | 35
  BOR by Investigator: Stable Disease | 56
  BOR by Investigator: Progressive Disease | 11
  BOR by Investigator: Not Done | 6

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR is the percentage (%) of subjects with a BOR of CR, PR, or SD, evaluated by CT or MRI scans every 28 days.
  Results are based on both BICR and on Investigator assessment.
  RECIST (v1.1) response criteria were as follows:
  CR: disappearance of all target lesions. Any pathological lymph node (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease from baseline in the sum of diameters of all target lesions.
  SD: neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for PD, taking as reference the smallest sum of diameters while on study.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (FGFR fusions) (disclosed 22 June 2022).
  There are no additional efficacy endpoints to assess for Cohort 1, thus efficacy data were not re-analyzed for the final analysis.
  Due to early termination of the study, no formal efficacy analyses were performed for Cohorts 2 and 3.
Time Frame: as for outcome 3
Population: Full Analysis Set (FAS), defined as all subjects in Cohort 1 who had received at least one dose of infigratinib.
Measure: Number (95% Confidence Interval); unit: Percentage (%) with CR, PR, or SD
Arm/Group | Cohort 1: FGFR2 Fusion/Rearrangements
Number analyzed (Participants) | 108
Percentage (%) with CR, PR, or SD
  DCR by BICR | 84.3 [76.0 to 90.6]
  DCR by Investigator | 84.3 [76.0 to 90.6]

5. Secondary Outcome: Progression-Free Survival (PFS)
Description: PFS was calculated as the number of months from the first dose of study drug to the first documented progression or death due to any cause, whichever occurred earlier. Subjects without an assessment of progression or death were censored at the last adequate tumor assessment. For subjects who had an event after ≥2 missed visits, the subject was censored at the last adequate tumor assessment before the missing visit.
  Disease progression was assessed per RECIST (v1.1) and defined as at least a 20% increase in the sum of diameters of all target lesions from that of the smallest sum on study and an absolute increase in target lesion of at least 5mm.
  Results are based on both BICR and on Investigator assessment.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (FGFR fusions) (disclosed 22 June 2022).
  Due to early termination of the study, no formal efficacy analyses were performed for Cohorts 2 and 3.
Time Frame: as for outcome 3
Population: Full Analysis Set (FAS), defined as all subjects in Cohort 1 who had received at least one dose of infigratinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: FGFR2 Fusion/Rearrangements
Number analyzed (Participants) | 108
months
  PFS by BICR | 7.29 [5.59 to 7.56]
  PFS by Investigator | 6.74 [5.55 to 7.56]

6. Secondary Outcome: Overall Survival (OS)
Description: OS was defined as the time (months) from the date of start of treatment to the date of death due to any cause.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (FGFR fusions) (disclosed 22 June 2022).
  Due to early termination of the study, no formal efficacy analyses were performed for Cohorts 2 and 3.
Time Frame: as for outcome 3
Population: Full Analysis Set (FAS), defined as all subjects in Cohort 1 who had received at least one dose of infigratinib.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: FGFR2 Fusion/Rearrangements
Number analyzed (Participants) | 108
months | 11.86 [10.68 to 14.85]

7. Secondary Outcome: Duration of Response (DOR)
Description: DOR is defined as the time (months) from the initial response to the time of the event; defined as the first documented progression or death due to any cause, whichever was earlier.
  Note that results are based on a subgroup of subjects with confirmed responses (CR or PR) as assessed by BICR or by the Investigator.
  RECIST (v1.1) response criteria was as follows:
  CR: disappearance of all target lesions. Any pathological lymph node (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease from baseline in the sum of diameters of all target lesions.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (FGFR fusions) (disclosed 22 June 2022).
  Due to early termination of the study, no formal efficacy analyses were performed for Cohorts 2 and 3.
Time Frame: as for outcome 3
Population: Full Analysis Set (FAS), defined as all subjects in Cohort 1 who had received at least one dose of infigratinib. Conducted in a subgroup of subjects who were confirmed responders (CR or PR) as assessed by BICR (N = 25) or by the Investigator (N = 35).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: FGFR2 Fusion/Rearrangements
Number analyzed (Participants) | 35
months
  DOR by BICR: number analyzed (Participants) | 25
  DOR by BICR | 5.55 [3.78 to 7.66]
  DOR by Investigator | 7.23 [5.16 to 9.00]

8. Secondary Outcome: Response Onset
Description: Response onset was defined as the time (months) from the first study treatment administration date to the initial response.
  Note that results are based on a subgroup of subjects with confirmed responses (CR or PR) as assessed by BICR or by the Investigator.
  RECIST (v1.1) response criteria was as follows:
  CR: disappearance of all target lesions. Any pathological lymph node (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease from baseline in the sum of diameters of all target lesions.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (FGFR fusions) (disclosed 22 June 2022).
  Due to early termination of the study, no formal efficacy analyses were performed for Cohorts 2 and 3.
Time Frame: as for outcome 3
Population: as for outcome 7
Measure: Median (Full Range); unit: months
Arm/Group | Cohort 1: FGFR2 Fusion/Rearrangements
Number analyzed (Participants) | 35
months
  Response onset by BICR: number analyzed (Participants) | 25
  Response onset by BICR | 3.61 [1.38 to 7.36]
  Response onset by Investigator | 1.94 [1.38 to 18.76]

9. Other Pre Specified Outcome: Growth Modulation Index (GMI)
Description: The GMI is defined as the ratio of PFS (months) during treatment with infigratinib relative to the time (months) to progression (TTP) during treatment with last prior line of therapy.
  Subjects served as their own control.
  Results are provided for both BICR and Investigator assessment.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (FGFR fusions) (disclosed 22 June 2022).
  Due to early termination of the study, no formal efficacy analyses were performed for Cohorts 2 and 3.
Time Frame: as for outcome 3
Population: Full Analysis Set (FAS), defined as all subjects in Cohort 1 who had received at least one dose of infigratinib. Conducted in a subgroup of subjects with both a PFS measure while on infigratinib and available TTP for their last prior line of therapy (N = 103).
Measure: Median (Full Range); unit: Ratio (PFS/TTP) in Months
Arm/Group | Cohort 1: FGFR2 Fusion/Rearrangements
Number analyzed (Participants) | 103
Ratio (PFS/TTP) in Months
  PFS by BICR | 1.22 [0.00 to 120]
  PFS by Investigator | 1.24 [0.00 to 120]

10. Post Hoc Outcome: Retrospective Analysis of Post-second-line Antineoplastic Treatment Outcomes on ORR
Description: Post-hoc subgroup assessment of efficacy in those subjects who were receiving infigratinib as a third or later line of treatment.
  Investigator-assessed ORR was obtained from subjects' medical histories to provide a baseline evaluation of their response after historical second-line antineoplastic treatment prior to infigratinib treatment. Investigator-assessed ORR was then calculated in the same subjects after third- or later-line infigratinib therapy.
  ORR is defined as the percentage (%) of patients with CR or PR, per RECIST (v1.1).
  RECIST (v1.1) response criteria were as follows:
  CR: disappearance of all target lesions. Any pathological lymph node (whether target or non-target) must have reduction in short axis to <10 mm.
  PR: at least a 30% decrease from baseline in the sum of diameters of all target lesions.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (22 June 2022).
  No formal efficacy analyses were performed for Cohorts 2 and 3.
Time Frame: as for outcome 3
Population: Full Analysis Set (FAS), defined as all subjects in Cohort 1 who had received at least one dose of infigratinib Conducted in a subgroup of subjects who were receiving infigratinib as a third or later line of treatment (N = 59).
Measure: Number (95% Confidence Interval); unit: Percentage (%) of patients with CR or PR
Arm/Group | Cohort 1: FGFR2 Fusion/Rearrangements
Number analyzed (Participants) | 59
Percentage (%) of patients with CR or PR
  After Second-Line Therapy (Prior to Infigratinib Treatment) | 0 [0.0 to 6.1]
  Third or Later-Line Therapy (Infigratinib) | 28.8 [17.8 to 42.1]

11. Post Hoc Outcome: Retrospective Analysis of Post-second-line Antineoplastic Treatment Outcomes on PFS
Description: Post-hoc subgroup assessment of efficacy in those subjects who were receiving infigratinib as a third or later line of treatment.
  Investigator-assessed PFS was obtained from subjects' medical histories to provide a baseline evaluation of their response after historical second-line antineoplastic treatment prior to infigratinib treatment. Investigator-assessed PFS was then calculated in the same subjects after third- or later-line infigratinib therapy.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (FGFR fusions) (disclosed 22 June 2022).
  Due to early termination of the study, no formal efficacy analyses were performed for Cohorts 2 and 3.
Time Frame: as for outcome 3
Population: Full Analysis Set (FAS), defined as all subjects in Cohort 1 who had received at least one dose of infigratinib. Conducted in a subgroup of subjects who were receiving infigratinib as a third or later line of treatment (N=59).
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Cohort 1: FGFR2 Fusion/Rearrangements
Number analyzed (Participants) | 59
months
  After Second-Line Therapy (Prior to Infigratinib Treatment) | 5.36 [3.25 to 8.15]
  Third or Later-Line Therapy (Infigratinib) | 6.93 [4.76 to 7.59]

12. Post Hoc Outcome: Retrospective Analysis of Post-second-line Antineoplastic Treatment Outcomes on BOR
Description: Post-hoc subgroup assessment of efficacy in those subjects who were receiving infigratinib as a third or later line of treatment.
  Investigator-assessed BOR was obtained from subjects' medical histories to provide a baseline evaluation of their response after historical second-line antineoplastic treatment prior to infigratinib treatment. Investigator-assessed BOR was then calculated in the same subjects after third- or later-line infigratinib therapy.
  The endpoint is summarized for the rate of BOR of PD, SD, PR, and CR.
  Note: The primary efficacy outcome measures were prespecified only for Cohort 1 (FGFR fusions) (disclosed 22 June 2022).
  Due to early termination of the study, no formal efficacy analyses were performed for Cohorts 2 and 3.
Time Frame: as for outcome 3
Population: Full Analysis Set (FAS), defined as all subjects in Cohort 1 who had received at least one dose of infigratinib Conducted in a subgroup of subjects who were receiving infigratinib as a third or later line of treatment (N=59).
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: FGFR2 Fusion/Rearrangements
Number analyzed (Participants) | 59
Participants
  After Second-Line Therapy (Prior to Infigratinib Treatment): Complete response | 0
  After Second-Line Therapy (Prior to Infigratinib Treatment): Partial response | 0
  After Second-Line Therapy (Prior to Infigratinib Treatment): Stable disease | 19
  After Second-Line Therapy (Prior to Infigratinib Treatment): Progressive disease | 22
  After Second-Line Therapy (Prior to Infigratinib Treatment): Unknown | 18
  After Second-Line Therapy (Prior to Infigratinib Treatment): Not done | 0
  Third or Later-Line Therapy (Infigratinib): Complete response | 0
  Third or Later-Line Therapy (Infigratinib): Partial response | 17
  Third or Later-Line Therapy (Infigratinib): Stable disease | 31
  Third or Later-Line Therapy (Infigratinib): Progressive disease | 7
  Third or Later-Line Therapy (Infigratinib): Unknown | 0
  Third or Later-Line Therapy (Infigratinib): Not done | 4

ADVERSE EVENTS:
Time Frame: From first administration of infigratinib with follow-up of at least 10 months after initial exposure. Data cutoff for Cohort 1 (primary analysis population) was 01 March 2021 (disclosed 22 June 2022). Data cutoff for Cohorts 2 and 3 (exploratory analysis only) was 07 February 2022.
Description: Adverse events (AEs) were assessed by the investigator according to CTCAE v4.03 and coded using MedDRA v21.0.
  Unless otherwise specified, treatment-emergent AEs are reported. AEs were considered treatment-emergent if they occurred on or after the first dose through the date of last dose +30 days.
Arm/Group | Cohort 1: FGFR2 Fusions | Cohort 2: Other FGFR Genetic Alterations | Cohort 3: FGFR2 Fusions and Prior FGFR Inhibitor
All-Cause Mortality (participants affected / at risk) | 93/108 | 19/25 | 7/10
Serious Adverse Events (participants affected / at risk) | 35/108 | 11/25 | 2/10
Other Adverse Events (participants affected / at risk) | 107/108 | 25/25 | 10/10
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: FGFR2 Fusions (N=108) | Cohort 2: Other FGFR Genetic Alterations (N=25) | Cohort 3: FGFR2 Fusions and Prior FGFR Inhibitor (N=10)
Anaemia (Blood and lymphatic system disorders) | 4 | 0 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0 | 0
Tachycardia (Cardiac disorders) | 1 | 0 | 0
Hypothyroidism (Endocrine disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 2 | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 0 | 0
Ascites (Gastrointestinal disorders) | 2 | 0 | 1
Constipation (Gastrointestinal disorders) | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0 | 0
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 1 | 0
Noninfective sialoadenitis (Gastrointestinal disorders) | 1 | 0 | 0
Pancreatitis (Gastrointestinal disorders) | 1 | 0 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 0 | 0
Intestinal ischaemia (Gastrointestinal disorders) | 0 | 1 | 0
Pyrexia (General disorders) | 4 | 2 | 0
Asthenia (General disorders) | 1 | 0 | 0
Gait disturbance (General disorders) | 1 | 0 | 0
General physical health deterioration (General disorders) | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 2 | 0 | 0
Bile duct obstruction (Hepatobiliary disorders) | 1 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 3 | 1 | 0
Cellulitis (Infections and infestations) | 2 | 0 | 0
Infection (Infections and infestations) | 2 | 0 | 0
Bacteraemia (Infections and infestations) | 1 | 0 | 0
Biliary abscess (Infections and infestations) | 1 | 0 | 0
Clostridium difficile colitis (Infections and infestations) | 1 | 0 | 0
Febrile infection (Infections and infestations) | 1 | 0 | 0
Intervertebral discitis (Infections and infestations) | 1 | 0 | 0
Lung infection (Infections and infestations) | 1 | 0 | 0
Peritonitis bacterial (Infections and infestations) | 1 | 0 | 0
Pneumonia (Infections and infestations) | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Stress fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Blood creatinine increased (Investigations) | 0 | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 4 | 0 | 0
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 0 | 1
Calciphylaxis (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Bone pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hepatic encephalopathy (Nervous system disorders) | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0
Acute kidney injury (Renal and urinary disorders) | 2 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 0 | 0
Pelvic pain (Reproductive system and breast disorders) | 1 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0
Peripheral ischaemia (Vascular disorders) | 0 | 1 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 0 | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 1
Device occlusion (Product Issues) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: FGFR2 Fusions (N=108) | Cohort 2: Other FGFR Genetic Alterations (N=25) | Cohort 3: FGFR2 Fusions and Prior FGFR Inhibitor (N=10)
Anaemia (Blood and lymphatic system disorders) | 20 | 5 | 0
Thrombocytopenia (Blood and lymphatic system disorders) | 9 | 2 | 0
Lymphopenia (Blood and lymphatic system disorders) | 7 | 1 | 0
Neutropenia (Blood and lymphatic system disorders) | 7 | 0 | 0
Dry eye (Eye disorders) | 39 | 3 | 4
Vision blurred (Eye disorders) | 23 | 4 | 1
Lacrimation increased (Eye disorders) | 13 | 2 | 0
Trichiasis (Eye disorders) | 13 | 4 | 0
Blepharitis (Eye disorders) | 12 | 2 | 0
Chorioretinopathy (Eye disorders) | 10 | 0 | 1
Punctate keratitis (Eye disorders) | 10 | 2 | 0
Cataract nuclear (Eye disorders) | 8 | 0 | 1
Growth of eyelashes (Eye disorders) | 7 | 0 | 0
Keratitis (Eye disorders) | 7 | 2 | 0
Ocular hyperaemia (Eye disorders) | 6 | 2 | 0
Subretinal fluid (Eye disorders) | 6 | 2 | 0
Visual acuity reduced (Eye disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 59 | 13 | 7
Constipation (Gastrointestinal disorders) | 34 | 11 | 3
Dry mouth (Gastrointestinal disorders) | 28 | 7 | 1
Diarrhoea (Gastrointestinal disorders) | 27 | 8 | 3
Vomiting (Gastrointestinal disorders) | 25 | 5 | 3
Nausea (Gastrointestinal disorders) | 21 | 10 | 3
Dyspepsia (Gastrointestinal disorders) | 20 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 19 | 2 | 1
Abdominal pain upper (Gastrointestinal disorders) | 16 | 4 | 0
Dysphagia (Gastrointestinal disorders) | 7 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 6 | 1 | 1
Oral pain (Gastrointestinal disorders) | 6 | 0 | 0
Abdominal discomfort (Gastrointestinal disorders) | 0 | 2 | 0
Abdominal pain lower (Gastrointestinal disorders) | 0 | 2 | 0
Oral dysaesthesia (Gastrointestinal disorders) | 0 | 2 | 0
Fatigue (General disorders) | 44 | 10 | 3
Pyrexia (General disorders) | 17 | 3 | 1
Oedema peripheral (General disorders) | 15 | 3 | 1
Chills (General disorders) | 8 | 1 | 0
Asthenia (General disorders) | 6 | 1 | 0
Non-cardiac chest pain (General disorders) | 6 | 0 | 0
Paronychia (Infections and infestations) | 11 | 2 | 0
Urinary tract infection (Infections and infestations) | 10 | 3 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 1
Blood creatinine increased (Investigations) | 27 | 8 | 1
Aspartate aminotransferase increased (Investigations) | 25 | 7 | 0
Alanine aminotransferase increased (Investigations) | 18 | 4 | 0
Blood alkaline phosphatase increased (Investigations) | 17 | 2 | 0
Weight decreased (Investigations) | 17 | 5 | 0
Lipase increased (Investigations) | 13 | 4 | 0
Blood bilirubin increased (Investigations) | 9 | 0 | 1
Amylase increased (Investigations) | 7 | 1 | 0
Gamma-glutamyltransferase increased (Investigations) | 1 | 2 | 0
Platelet count decreased (Investigations) | 0 | 2 | 0
Hyperphosphataemia (Metabolism and nutrition disorders) | 83 | 23 | 7
Hypercalcaemia (Metabolism and nutrition disorders) | 29 | 5 | 1
Decreased appetite (Metabolism and nutrition disorders) | 26 | 7 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 25 | 5 | 2
Hyponatraemia (Metabolism and nutrition disorders) | 14 | 2 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 9 | 1 | 0
Hypomagnesaemia (Metabolism and nutrition disorders) | 9 | 2 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 8 | 0 | 0
Hypokalaemia (Metabolism and nutrition disorders) | 8 | 2 | 0
Dehydration (Metabolism and nutrition disorders) | 7 | 2 | 0
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 7 | 1 | 0
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 2 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 4 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 17 | 5 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 16 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 14 | 4 | 0
Flank pain (Musculoskeletal and connective tissue disorders) | 7 | 0 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 7 | 2 | 0
Coccydynia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0
Dysgeusia (Nervous system disorders) | 34 | 6 | 0
Headache (Nervous system disorders) | 19 | 4 | 3
Dizziness (Nervous system disorders) | 10 | 3 | 0
Memory impairment (Nervous system disorders) | 6 | 0 | 0
Peripheral sensory neuropathy (Nervous system disorders) | 6 | 0 | 0
Insomnia (Psychiatric disorders) | 14 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 19 | 5 | 6
Cough (Respiratory, thoracic and mediastinal disorders) | 14 | 4 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 9 | 2 | 0
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 43 | 9 | 1
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 37 | 6 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 26 | 4 | 3
Nail discolouration (Skin and subcutaneous tissue disorders) | 20 | 4 | 2
Onychomadesis (Skin and subcutaneous tissue disorders) | 19 | 2 | 0
Nail disorder (Skin and subcutaneous tissue disorders) | 17 | 3 | 0
Onychalgia (Skin and subcutaneous tissue disorders) | 14 | 1 | 0
Onycholysis (Skin and subcutaneous tissue disorders) | 14 | 4 | 2
Nail ridging (Skin and subcutaneous tissue disorders) | 8 | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 8 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 7 | 0 | 2
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 6 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 0
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 3 | 0
Cataract (Eye disorders) | 0 | 1 | 1
Eye pain (Eye disorders) | 0 | 2 | 1
Keratopathy (Eye disorders) | 0 | 0 | 1
Retinal drusen (Eye disorders) | 0 | 0 | 1
Trichomegaly (Eye disorders) | 0 | 2 | 0
vitreous detachment (Eye disorders) | 0 | 0 | 1
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 1
Ascites (Gastrointestinal disorders) | 0 | 0 | 1
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Retching (Gastrointestinal disorders) | 0 | 0 | 1
Enterocolitis infectious (Infections and infestations) | 0 | 0 | 1
Infection (Infections and infestations) | 0 | 0 | 1
Vulvovaginal candidiasis (Infections and infestations) | 0 | 0 | 1
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Creatinine renal clearance decreased (Investigations) | 0 | 0 | 1
Pain in jaw (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 0 | 0 | 1
Chromaturia (Renal and urinary disorders) | 0 | 0 | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 1
Skin exfoliation (Skin and subcutaneous tissue disorders) | 0 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2020-01-15): https://cdn.clinicaltrials.gov/large-docs/67/NCT02150967/Prot_000.pdf
  • Statistical Analysis Plan (2020-05-13): https://cdn.clinicaltrials.gov/large-docs/67/NCT02150967/SAP_001.pdf